CLINICAL TRIAL: NCT03111693
Title: CT Evaluation of Cardiovascular Risk Markers in Obese Patients
Acronym: RisqOScan
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-312; 2014-A00975-42 (Other: 2014-A00975-42)
Record Dates: First submitted 2017-03-30; First posted 2017-04-13 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Epicardial Fat; Obesity; Cardiovascular Risks Markers; Metabolic Syndrome; Low Dose Computed Tomography
Keywords: Epicardial fat; Obesity; Cardiovascular risks markers; Metabolic syndrome; Low dose computed tomography
MeSH Terms: conditions — Obesity; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- obese patients: obese patients of our clinical nutrition service, hospitalized for nutrional assessement, are included.
  Interventions: Other: Unenhanced Coro-CT

INTERVENTIONS:
Other: Unenhanced Coro-CT — All unenhanced coroCT examinations are performed on the same 64-Row CT scanner (discovery CT 750 HD scanner, GE Helthcare), using prospective ECG-triggerring.

SUMMARY:
Obesity is a chronic metabolic disorder : it leads to coronary heart disease and early atherosclerosis.

Coronary artery calcium measured by CT is known as a robust predictor to predict risk for cardiac events in symptomatic and asymptomatic individuals. Furthermore, recent studies show that other CT risk factor exists, independent of calcium scoring, such as epicardial fat, intrathoracic fat and visceral fat.

The aim of this prospective study is to evaluate these new cardiovascular risk markers in obese patients, using standard dose CT and low dose CT with adaptative statistical iterative reconstruction.

DETAILED DESCRIPTION:
In this prospective single-center study, obese patients of our clinical nutrition service, hospitalized for nutritional assessement, are included.

All unenhanced coroCT examinations are performed on the same 64-Row CT scanner (discovery CT 750 HD scanner, GE Healthcare), using prospective ECG-triggerring. The investigation protocol began with a standard-dose acquisition followed immediately by a low-dose acquisition, recorded over strictly identical segments (identical first and last sections).

After these two examinations, estimated dose values are less than the diagnostic scan reference level for a coroCT.

ELIGIBILITY:
Inclusion Criteria:

* obesity >30 indicated non enhanced coroCT for calcium scoring.

Exclusion Criteria:

* <18 ans
* low Framingham scoring
* pregnancy
* not providing informed consent
* history of cardiovascular disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: obese population
Sampling Method: Non-Probability Sample
Enrollment: 123 (Estimated)
Dates: Start 2014-11 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Epicardial fat evaluation in obese population | at day 1

SECONDARY OUTCOMES:
Calcium scoring evaluation | at day 1

CONTACTS AND LOCATIONS:
Overall Officials: Lucie CASSAGNES, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France